CLINICAL TRIAL: NCT00316472
Title: The Effect of Oral Niacinamide on Serum Phosphorus Levels in Hemodialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Daniel Coyne, MD, Washington University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC05-0958
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Hyperphosphatemia
Keywords: Hyperphosphatemia; End Stage Renal Disease; Renal Osteodystrophy
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Niacinamide

INTERVENTIONS:
Drug: Niacinamide

SUMMARY:
Elevated phosphorus levels are a common problem in dialysis patients. However, it is associated with an increase in death and hospitalizations. Current treatment is comprised of dietary modifications and phosphorus binders - though this is often not enough for many of our patients. Our trial investigates the use of niacinamide, a form of vitamin B, in decreasing serum phosphorus levels.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled crossover study comparing niacinamide versus placebo in the reduction of serum phosphorus in hemodialysis patients. A determination of baseline laboratory values (serum phosphorus, calcium, albumin, biPTH, uric acid, complete blood count (CBC), and an NMR lipid panel) will precede the administration of the study drugs. The study will span a period of 21 weeks during which phosphorus levels will be checked on a weekly basis. Phosphorus binder dose will remain unchanged unless for safety reasons. For the first 8 weeks of treatment, patients will be randomized to either placebo or niacinamide. Both medications will be administered with a starting dose of one capsule twice per day (BID). Niacinamide and placebo will be formulated in 250 mg capsules. Placebo will be packaged to resemble the study drug in all physical attributes. The dose of niacinamide or placebo will be increased to 500 mg (2 capsules) BID at week 3 and 750 mg (3 capsules) BID at week 5. If hypophosphatemia (< 3.5 mg/dl) is present, then titration will not occur and the previous dose will be continued. However, titration will resume in subsequent weeks if the serum phosphorus is greater than 3.5 mg/dl. After 8 weeks, patients will undergo a 2 week washout period, then crossover from treatment arm to placebo, or vice versa, at week 11.

At the beginning of week 11, patients will cross over to the other treatment arm (either placebo or niacinamide) at one capsule (250 mg) twice per day. Subsequent titration will occur at week 13 and week 15. The treatment phase will be completed at the end of week 18. A set of labs will be drawn at the start of week 19, followed by a two week washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Capable of giving informed consent
3. Duration of chronic hemodialysis > 90 days
4. Dose of phosphorus binder(s) stable over previous 2 week period
5. Serum Phosphorus > 4.9 mg/dL based on most recent laboratory data within 1 month of enrollment

Exclusion Criteria:

1. Pregnancy
2. Known liver disease
3. Active peptic ulcer disease
4. Treatment with carbamazepine
5. Intolerance to niacinamide
6. Current medication regimen including niacin or niacinamide-containing vitamins
7. More than 1 missed hemodialysis session in the last 30 days
8. Planned or expected surgical procedure in the next 4 months
9. Patients in nursing homes or extended care facilities where administration of the study drug may not be appropriately given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint: The change in serum phosphorus after 8 weeks of niacinamide versus placebo.

SECONDARY OUTCOMES:
Secondary endpoints: To assess the effects of niacinamide on calcium-phosphorus product, biointact parathyroid hormone levels (biPTH), and lipid profiles after 8 weeks of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Coyne, M.D>, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Result] Cheng SC, Young DO, Huang Y, Delmez JA, Coyne DW. A randomized, double-blind, placebo-controlled trial of niacinamide for reduction of phosphorus in hemodialysis patients. Clin J Am Soc Nephrol. 2008 Jul;3(4):1131-8. doi: 10.2215/CJN.04211007. Epub 2008 Apr 2. PMID 18385391
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086